CLINICAL TRIAL: NCT04475809
Title: Different Maneuvers for Reducing Post-laparoscopic Shoulder and Abdominal Pain: A Randomized Controlled Trial
Brief Title: Different Maneuvers for Reducing Post-laparoscopic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Shereen Elsayed Abd Ellatif, lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6251-1207-2020
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Gynecologic Disease
Keywords: Pulmonary recruitment maneuvers; low-pressure pneumoperitoneum; laparoscopic Shoulder and Abdominal Pain; laparoscopic gynecologic surgery; intraperitoneal saline infusion
MeSH Terms: conditions — Genital Diseases, Female; Abdominal Pain

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into two equal groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) double-blinded ( patient and outcome assessors)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group C (Placebo Comparator): high intra-abdominal pressure
  Interventions: Procedure: group C
- Group L (Active Comparator): low intra-abdominal pressure
  Interventions: Procedure: Group L
- Group LR (Active Comparator): low intra-abdominal pressure with pulmonary recruitment maneuver group
  Interventions: Procedure: Group LR
- Group LS (Active Comparator): low intra-abdominal pressure with intraperitoneal saline infusion group
  Interventions: Procedure: Group LS

INTERVENTIONS:
Procedure: group C — laparoscopy will be performed with 14-16 mmHg intra-abdominal pressure. At the end of the procedure routine method for CO2 removal, passive exsufflation, will be used by applying gentle abdominal pressure to evacuate the residual gas through the port site.
  Arms: Group C
Procedure: Group L — laparoscopy will be performed with 8-10 mmHg intra-abdominal pressure and routine passive exsufflation will be applied for CO2 removal at the end of the procedure.
  Arms: Group L
Procedure: Group LR — the intra-abdominal pressure will be kept at 8-10 mmHg during laparoscopy. At the end of the procedure pulmonary recruitment maneuver (PRM) will be done; which consists of five manual pulmonary inflations at a maximum pressure of 40 cm H2O and the fifth will be held for 5 seconds. During this procedure, the surgeon is instructed to keep the port sleeve valve fully opened to allow the CO2 to escape the abdominal cavity.
  Arms: Group LR
Procedure: Group LS — the intra-abdominal pressure will be kept at 8-10 mmHg during laparoscopy. At the end of the procedure, intraperitoneal normal saline (IPS) will be infused for removal of the intra-abdominal CO2; in which we fill the upper part of the abdominal cavity evenly and bilaterally with isotonic normal saline (15-20 mL/kg body weight)
  Arms: Group LS

SUMMARY:
* Laparoscopic surgeries are becoming more attractive because of early recovery. However, post-laparoscopic shoulder and upper abdominal pain may cause more discomfort to the patient than the pain at the incision site
* Many strategies have been attempted, such as the use of nonsteroidal anti-inflammatory drugs; however, the effect is limited, and there are no reliable methods available yet.
* Recently, some techniques are introduced that can potentially alleviate various types of pain through different mechanisms in patients after laparoscopic surgery such as low-pressure pneumoperitoneum, intraperitoneal normal saline infusion, and pulmonary recruitment maneuvers.
* the investigators conduct this randomized controlled trial to evaluate the effectiveness of different strategies on reducing the intensity of post-laparoscopic shoulder and abdominal pain in patients undergoing laparoscopic gynecologic surgeries.

DETAILED DESCRIPTION:
Laparoscopic surgery is becoming more popular due to smaller incision, faster recovery, less postoperative pain, and earlier returns to normal activity . However post-laparoscopic shoulder and upper abdominal pain may upset the patient more than the pain at the incision site. The incidence of shoulder pain after laparoscopic gynecological surgery varies from 35% to 80% and could be so severe at 24 hours after laparoscopic hysterectomy as well.

The mechanism of post laparoscopic shoulder and abdominal pain attributes to the insufflated co2 in the abdominal cavity and become entrapped between the liver and the right diaphragm causing irritation of the phrenic nerve, diaphragm and referred pain in the C4 dermatome. On the other hand, the prolonged exposure to residual CO2 dissolution leads to intra-abdominal acidosis and consequent peritoneal irritation and abdominal pain.

As long as the retention of CO2 is the key factor in the laparoscopy-induced shoulder and abdominal pain, many strategies have been evolved to alleviate different types of pain in patients undergoing laparoscopic surgeries such as usage of low-pressure pneumoperitoneum (8-10 mmHg) that result in reducing the intensity of postoperative pain in comparison to standard high-pressure pneumoperitoneum (12-15 mmHg). Although this low pressure may impair visualization and jeopardize the surgeon's comfort during surgery, this method is proven to be safe and feasible.

One of the maneuvers that have been proposed is an intraperitoneal normal saline infusion (IPS) that increases intraperitoneal pressure to enhance the removal of residual CO2, as well as offers a physiologic buffer system to wash out excess CO2.

Pulmonary recruitment maneuvers (PRM) has also a potential beneficial effect on alleviating post-laparoscopic pain by mechanically increasing intraperitoneal pressure to accelerate the elimination of residual CO2.

Because these variable techniques are mediated through different mechanisms, the investigators hypothesize that combination of two different maneuvers may be ideal and more effective in reducing post-laparoscopic shoulder and abdominal pain than any single or standard maneuver in patients undergoing laparoscopic gynecologic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* BMI ≤35 kg/m2.
* ASA I and ASA II.
* Scheduled for elective laparoscopic gynecologic surgeries for benign lesions under general anesthesia.

Exclusion Criteria:

* Patients with pre-existing chronic pain disorders.
* Patients on opioid or sedative use.
* Psychological and mental disorders.
* Severe hypertensive, cardiac, hepatic and renal patients.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
changes in assessment of shoulder, abdominal and incisional pain | at 1, 2, 4, 6, 12, 24, 48,72,96 hours postoperatively
  will be assessed by visual analogue scale (VAS) scale, On a scale of 0-10, the patient will learn to quantify postoperative pain where 0= No pain and 10= Maximum worst pain.

SECONDARY OUTCOMES:
Time of first request of analgesia | within 24 hour postoperative
  time elapsed from patient arrival to post anesthesia care unit to time of first patient call for analgesia
Total rescue analgesic requirement | during the first postoperative 96 hours
  if VAS ≥3 or on patient request, rescue analgesia will be given

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, zagazig university, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Background] Kaloo P, Armstrong S, Kaloo C, Jordan V. Interventions to reduce shoulder pain following gynaecological laparoscopic procedures. Cochrane Database Syst Rev. 2019 Jan 30;1(1):CD011101. doi: 10.1002/14651858.CD011101.pub2. PMID 30699235
- [Background] Tsai HW, Chen YJ, Ho CM, Hseu SS, Chao KC, Tsai SK, Wang PH. Maneuvers to decrease laparoscopy-induced shoulder and upper abdominal pain: a randomized controlled study. Arch Surg. 2011 Dec;146(12):1360-6. doi: 10.1001/archsurg.2011.597. PMID 22184293
- [Background] Yasir M, Mehta KS, Banday VH, Aiman A, Masood I, Iqbal B. Evaluation of post operative shoulder tip pain in low pressure versus standard pressure pneumoperitoneum during laparoscopic cholecystectomy. Surgeon. 2012 Apr;10(2):71-4. doi: 10.1016/j.surge.2011.02.003. Epub 2011 Mar 21. PMID 22385527
- [Background] Pergialiotis V, Vlachos DE, Kontzoglou K, Perrea D, Vlachos GD. Pulmonary recruitment maneuver to reduce pain after laparoscopy: a meta-analysis of randomized controlled trials. Surg Endosc. 2015 Aug;29(8):2101-8. doi: 10.1007/s00464-014-3934-7. Epub 2014 Nov 1. PMID 25361653
- [Background] Davari-Tanha F, Samimi S, Khalaj Z, Bastanhagh E. Comparison of Intraperitoneal Normal Saline Infusion with Pulmonary Recruitment Maneuver in Reducing Shoulder and Upper Abdomen Pain Following Gynecologic Laparoscopic Procedures: A Randomized, Controlled, Triple-Blind Trial. Anesth Pain Med. 2019 Jun 2;9(3):e92444. doi: 10.5812/aapm.92444. eCollection 2019 Jun. PMID 31497525
- [Background] Sharami SH, Sharami MB, Abdollahzadeh M, Keyvan A. Randomised clinical trial of the influence of pulmonary recruitment manoeuvre on reducing shoulder pain after laparoscopy. J Obstet Gynaecol. 2010;30(5):505-10. doi: 10.3109/01443611003802313. PMID 20604657